CLINICAL TRIAL: NCT03644966
Title: Probiotic and Effects on Multi-Drug Resistant Urinary Tract Infection
Brief Title: Probiotics and Multi-Drug Resistant Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017564
Record Dates: First submitted 2018-08-06; First posted 2018-08-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Urinary Tract Infections; Recurrent UTI; Antibiotic Resistant Infection
Keywords: Probiotics; multi-drug resistant UTI; recurrent UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic + Antibiotic (Experimental): 50 subjects to receive probiotic supplement once daily for 6 months in capsule form, in addition to standard antibiotic regimen for treatment of UTI.
  Interventions: Dietary Supplement: Bifidobacterium infantis; Drug: Antibiotics
- Placebo + Antibiotic (Active Comparator): 50 subjects to receive placebo once daily for 6 months in capsule form, in addition to antibiotic regimen for treatment of UTI.
  Interventions: Other: Placebo; Drug: Antibiotics

INTERVENTIONS:
Dietary Supplement: Bifidobacterium infantis — Probiotics
  Other Names: Align
  Arms: Probiotic + Antibiotic
Other: Placebo — Sugar pill manufactured to mimic probiotic tablet
  Other Names: Placebo (for Probiotic)
  Arms: Placebo + Antibiotic
Drug: Antibiotics — Per Infectious Disease Society guidelines for Antimicrobial treatment of uncomplicated cystitis and pyelonephritis in women

SUMMARY:
This pilot study is a single-site randomized, double blinded placebo-controlled in females with recurrent multi-drug resistant (MDR) urinary tract infections(UTI). Our study hypothesizes that a novel probiotic strain improves antibiotic sensitivity patterns in these former MDR UTIs.

DETAILED DESCRIPTION:
The aims of this study are (1) to evaluate the effects of six months of probiotic therapy in addition to standard of care in changing sensitivity patterns of MDR bacteria causing recurrent UTI, (2) analyze the genetic composition of MDR bacterial isolates causing recurrent UTI before and after administration of probiotic vs. placebo, with standard of care antibiotics.

Study subjects will be asked to take a either a probiotic supplement or placebo at a dose of 1 caplet per day for 24 weeks in addition to antibiotic regimen. Subjects will be followed for 12 months. The outcome measure is the percent of probiotic ingestors vs placebo ingestors who experience a change in antibiotic susceptibility over this time period. The secondary outcome measure is the evaluation of genetic composition of bacteria recurring after probiotic vs. placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-90
* Ability to void spontaneously
* Suffers from recurrent multi-drug resistant or extensively drug resistant urinary tract infections caused by E.coli, Klebsiella, Enterococcus, Citrobacter, Proteus, Enterobacter, Serratia and Providencia.

Exclusion Criteria:

* Has staghorn renal calculi, chronic hydronephrosis, intermittent catherization, indwelling urinary catheters, urinary diversions, end stage renal disease on hemodialysis, transplantation, HIV, cirrhosis, pancreatitis, allergy to soy or milk/milk proteins or lactose intolerance
* Pregnant or breastfeeding
* Currently taking probiotics. 4 week washout.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Resistance Pattern | 6-8 weeks after initial dose
  The change in the quantity of antibiotics reported to be resistant per organism per culture per patient.
Bacterial isolate genomic characteristics | 12 months after initial dose
  genomic sequencing of bacterial isolates to determine genetic identity

SECONDARY OUTCOMES:
UTI reduction | 12 months after initial dose
  The quantity of reduction of all urinary tract infections (UTI) in treatment arm vs. placebo from baseline.
Antibiotics Quantity | 12 months after initial dose
  The quantity of antibiotics prescribed in treatment arm vs. placebo.
Healthcare visit | 12 months after initial dose
  The quantity of ER visits/urgent care visits/hospitalizations/outpatient clinic visits in treatment arm vs. placebo.
Length of time for change in resistance | 12 months after initial dose
  The amount of time it takes to note changes in antibiotic sensitivity patterns while on the treatment arm.
Sensitivity pattern post-probiotic therapy | 12 months after initial dose
  The change in the quantity of antibiotics reported to be resistant per organism

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Health System, Jefferson, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naderi A, Kasra-Kermanshahi R, Gharavi S, Imani Fooladi AA, Abdollahpour Alitappeh M, Saffarian P. Study of antagonistic effects of Lactobacillus strains as probiotics on multi drug resistant (MDR) bacteria isolated from urinary tract infections (UTIs). Iran J Basic Med Sci. 2014 Mar;17(3):201-8. PMID 24847423
- [Background] Schwenger EM, Tejani AM, Loewen PS. Probiotics for preventing urinary tract infections in adults and children. Cochrane Database Syst Rev. 2015 Dec 23;2015(12):CD008772. doi: 10.1002/14651858.CD008772.pub2. PMID 26695595
- [Background] Simmering JE, Tang F, Cavanaugh JE, Polgreen LA, Polgreen PM. The Increase in Hospitalizations for Urinary Tract Infections and the Associated Costs in the United States, 1998-2011. Open Forum Infect Dis. 2017 Feb 24;4(1):ofw281. doi: 10.1093/ofid/ofw281. eCollection 2017 Winter. PMID 28480273
- [Background] Barclay J, Veeratterapillay R, Harding C. Non-antibiotic options for recurrent urinary tract infections in women. BMJ. 2017 Nov 23;359:j5193. doi: 10.1136/bmj.j5193. No abstract available. PMID 29170359
- [Background] Vahedi-Shahandashti R, Kasra-Kermanshahi R, Shokouhfard M, Ghadam P, Feizabadi MM, Teimourian S. Antagonistic activities of some probiotic lactobacilli culture supernatant on Serratia marcescens swarming motility and antibiotic resistance. Iran J Microbiol. 2017 Dec;9(6):348-355. PMID 29487733
- [Background] Lau CS, Chamberlain RS. Probiotics are effective at preventing Clostridium difficile-associated diarrhea: a systematic review and meta-analysis. Int J Gen Med. 2016 Feb 22;9:27-37. doi: 10.2147/IJGM.S98280. eCollection 2016. PMID 26955289
- [Background] Favier C, Neut C, Mizon C, Cortot A, Colombel JF, Mizon J. Fecal beta-D-galactosidase production and Bifidobacteria are decreased in Crohn's disease. Dig Dis Sci. 1997 Apr;42(4):817-22. doi: 10.1023/a:1018876400528. PMID 9125655
- [Background] Gupta K, Hooton TM, Naber KG, Wullt B, Colgan R, Miller LG, Moran GJ, Nicolle LE, Raz R, Schaeffer AJ, Soper DE; Infectious Diseases Society of America; European Society for Microbiology and Infectious Diseases. International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women: A 2010 update by the Infectious Diseases Society of America and the European Society for Microbiology and Infectious Diseases. Clin Infect Dis. 2011 Mar 1;52(5):e103-20. doi: 10.1093/cid/ciq257. PMID 21292654